CLINICAL TRIAL: NCT01615510
Title: Evaluation of the Antihyperalgesic Effect of Tapentadol in Two Human Experimental Models of: 1) Cold and Mechanical Hyperalgesia Evoked by Topical High-concentration Menthol , 2) Heat and Mechanical Hyperalgesia by Capsaicin.
Brief Title: Evaluation of the Antihyperalgesic Effect of Tapentadol in Two Human Experimental Models
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Ralf Baron, Professor Dr., head of division of neurological pain research and therapy, University Hospital Schleswig-Holstein
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: TapCapMentho01
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Pain; Hyperalgesia; Allodynia
MeSH Terms: conditions — Pain; Hyperalgesia | interventions — Tapentadol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Capsaicin (topical) (Experimental): 300 µL of 0.6% capsaicin in 45% ethanol, topically applied on the forearm intervention: tapentadol immediate release or placebo
  Interventions: Drug: Tapentadol immediate release; Drug: placebo
- Menthol (topical) (Experimental): 1000 µL of 40% menthol in 90% ethanol, topically applied on the forearm intervention: tapentadol immediate release or placebo
  Interventions: Drug: Tapentadol immediate release; Drug: placebo

INTERVENTIONS:
Drug: Tapentadol immediate release — 100 mg, single administration
  Other Names: Palexia IR
Drug: placebo — placebo, single administration
  Other Names: P Lichtenstein

SUMMARY:
MOR-NRI like Tapentadol are expected to reduce signs and symptoms of central sensitisation besides effectively reducing pain intensity in pain. Human pain surrogate models can serve in this proof-of-concept study to further elucidate this assumption.

DETAILED DESCRIPTION:
To evaluate exploratory the antihyperalgesic effect of a single dose of Palexia® IR (Tapentadol) in two human experimental models of 1) cold and mechanical (pinprick) hyperalgesia after topical application of menthol at high-concentration [40%] and 2) of heat and mechanical (pinprick) hyperalgesia by topical applied capsaicin [0.6%] in comparison to placebo. Therefore, cold, heat and mechanical hyperalgesia and allodynia will be determined by parameters of the Quantitative Sensory Testing (QST). These parameters are cold and heat pain thresholds, mechanical pain threshold and sensitivity as well as dynamic mechanical allodynia. Further, the areas of dynamic mechanical allodynia and pinprick-hyperalgesia will be determined at each timepoint of QST-assessement.

ELIGIBILITY:
Inclusion Criteria:

1. Provided written informed consent to participating in the trial.
2. Caucasian, female or male, and aged 18 years to 55 years, inclusive.
3. Body mass index between 18.5 kg/m2 and 30 kg/m2, inclusive, with a lower body weight limit of 50 kg.
4. In good health as determined by medical history, physical examination, 12-lead ECG, vital signs (pulse rate, respiratory rate, systolic and diastolic blood pressure), oxygen saturation, and laboratory monitoring (hematology, clinical chemistry, clotting, and urinalysis).
5. Subjects must be able to feel thermal and mechanical sensation (cold, warm, sharp, unpleasant sensation) on normal skin (at the forearm intended for menthol / capsaicin administration) confirmed by routine neurological bed-side testing.
6. Female subjects must be postmenopausal (with at least 2 years since last menstruation), surgically sterile (e.g., after hysterectomy or bilateral oophorectomy), or practicing an effective method of birth control (e.g., oral contraceptives, contraceptive injections, intrauterine device, double-barrier method, contraceptive patch, male partner sterilization) at the Enrollment Visit and during the trial.
7. Female subjects of childbearing potential must have a negative serum hCG test at the Enrollment Visit.

Exclusion Criteria:

1. The subject has received any of the IMPs or used an investigational medical device within 30 days or within a period less than 10 times the half life of an investigational drug, whichever is longer, before the first dose of IMP is scheduled.
2. History or presence of opioid abuse, drug abuse, or alcohol abuse or presence of an acute intoxication with alcohol, hypnotics, centrally acting analgesics, or psychotropic drugs.
3. Positive or missing drugs of abuse screening (alcohol breath test, urine screening test for drugs of abuse).
4. Diseases or conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
5. History or presence of severe respiratory depression with hypoxia and/or hypocapnia, severe chronic obstructive pulmonary disease, cor pulmonale, severe bronchial asthma, paralytic ileus.
6. History or presence of hypersensitivity to Tapentadol, menthol, capsaicin/chili peppers or any of the other excipients of the Palexia® IR (Tapentadol), menthol, or capsaicin formulations or to opioid antagonists (e.g., naloxone).
7. Subjects who have used any prescribed and non-prescribed systemic or topical medication, except contraceptives, on a daily base within 14 days before the Enrolment Visit, or anticipated use from the Enrolment Visit until the first administration of the IMP.
8. History or presence of seizure disorder and/or epilepsy or any condition associated with a significant risk for seizure disorder or epilepsy.
9. History of orthostatic hypotension.
10. Blood donation or acute loss of blood (more than 100 mL) during the 1 month before the enrollment visit, or intention to donate blood or blood products during the trial or within 1 month following the completion of the trial.
11. Pregnant or breastfeeding women.
12. Known or suspected of not being able to comply with procedures described in the trial protocol.
13. Not able to communicate meaningfully with the investigator and staff.
14. Preplanned surgery or procedures that would interfere with the conduct of the trial.
15. Acute skin disease, lesions, acute sunburn, extensive tattoos or scars at the forearm where the menthol / capsaicin application is planned.
16. Employee of the Investigator or trial site, with direct involvement in the proposed trial or other trials under the direction of that Investigator or trial site, as well as family members of the employees or the Investigator
17. Administration of a monoaminoxidase-inhibitor (MAO-Inhibitor) within 14 days prior to recruitment visit.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
QST parameters | period 1 - period 2 (approx. 18 days)
  The primary objective is to evaluate the antihyperalgesic effect of a single dose of Tapentadol immediate release (IR) in two human experimental models:
  1. cold pain threshold (menthol only),
  2. heat pain thresholds (capsaicin only),
  3. mechanical pain threshold
  4. mechanical pain sensitivity,
  5. dynamic mechanical allodynia,
  6. area of dynamic mechanical allodynia and
  7. area of pinprick-hyperalges

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Baron, Professor, Principal Investigator — Head of Division of Neurological Pain Research and Therapy
Locations (1):
- Department of Neurology, Kiel, Germany

REFERENCES:
- [Derived] Forster M, Helfert S, Dierschke R, Grosskopf M, Hullemann P, Keller T, Baron R, Binder A. Evaluation of the antihyperalgesic effect of tapentadol in two human evoked pain models - the TapCapMentho pilot trial. Expert Opin Pharmacother. 2016 Sep;17(13):1717-25. doi: 10.1080/14656566.2016.1201071. Epub 2016 Aug 10. PMID 27295489